CLINICAL TRIAL: NCT03196063
Title: Effectiveness of Two Exercise Protocols in the Treatment of Patients With Patellar Tendinopathy: a Randomized Controlled Trial
Brief Title: Effectiveness of Two Exercise Protocols in the Treatment of Patients With Patellar Tendinopathy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study stopped because we could not recruit patients in the available time
Sponsor: Universidade Cidade de Sao Paulo (Other)
Responsible Party: Principal Investigator, Cristina Maria Nunes Cabral, Professor, Universidade Cidade de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNICID16
Record Dates: First submitted 2017-06-20; First posted 2017-06-22 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Patellar Tendinopathy
Keywords: Exercise Therapy; Heavy Slow Resistance Program; Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eccentric (Active Comparator): Patients allocated in this group will perform three sets of 15 unipodal squats with the affected limb on an inclined plane. The patient will be instructed to perform only the eccentric phase of the exercise, keeping the torso erect and flexing the knee up to 90 degrees. The return to the initial position will be performed with the unaffected leg. To increase exercise load, the patient will carry a bag with washers. This protocol will last eight weeks, with 24 face-to-face sessions.
  Both groups will also receive a protocol with complementary isotonic exercises, focusing on the strengthening of gluteus maximus, gluteus medius, hamstrings and calves.
  Interventions: Other: Eccentric
- Modified protocol (Experimental): Patients allocated in this group will receive treatment based on a protocol published in a clinical practice guide, with modifications to make the protocol more pragmatic. Thus, the use of mechanotherapy devices will be replaced by free weight exercises, so that the protocol can be performed in environments that do not offer this type of machinery. This protocol is composed of four exercise stages, being the first three stages performed in the presence of the physiotherapist, and will last eight weeks with approximately 24 face-to-face sessions.
  Both groups will receive a protocol with complementary isotonic exercises, focusing on the strengthening of gluteus maximus, gluteus medius, hamstrings and calves.
  Interventions: Other: Modified Protocol

INTERVENTIONS:
Other: Eccentric — Exercises based on eccentric contractions of the quadriceps femoris muscle, using a 15º inclined plane. A serie of 15 repetitions of the squat will be performed, with the frequency of three times a week for eight weeks. The load of the exercises will be increased weekly.
  Other Names: Eccentric exercise
  Arms: Eccentric
Other: Modified Protocol — Protocol based on the Heavy Slow resistance program, with the addition of an isometric phase at the beginning of the protocol, and with exercises using body weight without the use of mechanotherapy.
  Other Names: Heavy Slow Resistance Program
  Arms: Modified protocol

SUMMARY:
Patellar tendinopathy is characterized by anterior pain in the knee, due to the great demand imposed on the extensor mechanism of the knee. Evidence shows that the most appropriate treatment for this condition is the conservative treatment, through strengthening with eccentric exercises. However, a recent editorial proposes a new treatment protocol based on concentric and eccentric exercises, with the initial prescription of isometric exercises. The hypothesis of this study is that the protocol is as good as the eccentric exercises, generating less pain.

ELIGIBILITY:
Inclusion Criteria:

* patients with chronic unilateral patellar tendinopathy confirmed by the reproduction of the pain during the palpation test in the region of the lower pole of the patella
* presence of pain for three months or more
* both genders
* body mass index less than 30 kg/m²
* age between 18 and 40 years
* practice of physical activity on a regular basis
* pain intensity ≥ 3 points on the pain numerical rating scale in the anterior region of the knee, specifically in the region of the lower pole of the patella when performing squatting, jumping or activities with change of direction
* score < 80 points on the Victorian Institute of Sport Assessment-Patella (VISA-P)
* blazine functional scale between 1 and 3

Exclusion Criteria:

* patients who have previous pain in the knee that does not correspond to patellar tendinopathy
* previous rupture of the patellar tendon (blazin functional scale at level 4)
* previous surgery or infiltration of the patellar tendon in the last six months
* inflammatory diseases
* diabetes mellitus
* lower limbs injuries
* other chronic pain conditions that prevent exercise, such as severe hip and knee osteoarthrosis and joint fractures.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Pain intensity during rest | 8 weeks after randomization
  This outcome will be evaluated by an 11-point scale ranging from 0 to 10, in which 0 represents "no pain" and 10 represents "pain as bad as it could be." The participant will classify his average pain in the last 7 days.
Functional capacity | 8 weeks after randomization
  VISA-P questionnaire assesses the symptoms and disability of patients with patellar tendinopathy. It is a questionnaire with eight questions, six of them on a Likert scale, ranging from 0 to 10 points, where 0 represents the maximum severity of the disease and 10 represents no pain or limitation. Question 7 has four possible answers (0, 4, 7 and 10 points). Question 8 has a subdivision (8A, 8B and 8C), in which only one can be answered, depending on the perception of pain during sport activities, varying up to 30 points. The total score of the questionnaire varies between 0 and 100 points, with 100 points corresponding to the absence of pain or disability.

SECONDARY OUTCOMES:
Pain intensity during rest | 12 weeks and 6 months after randomization
  This outcome will be evaluated by an 11-point scale ranging from 0 to 10, in which 0 represents "no pain" and 10 represents "pain as bad as it could be." The participant will classify his average pain in the last 7 days.
Functional capacity | 12 weeks and 6 months after randomization
  VISA-P questionnaire assesses the symptoms and disability of patients with patellar tendinopathy. It is a questionnaire with eight questions, six of them on a Likert scale, ranging from 0 to 10 points, where 0 represents the maximum severity of the disease and 10 represents no pain or limitation. Question 7 has four possible answers (0, 4, 7 and 10 points). Question 8 has a subdivision (8A, 8B and 8C), in which only one can be answered, depending on the perception of pain during sport activities, varying up to 30 points. The total score of the questionnaire varies between 0 and 100 points, with 100 points corresponding to the absence of pain or disability.
Pain intensity during squat | 8 weeks after randomization
  This outcome will be evaluated by an 11-point scale ranging from 0 to 10, in which 0 represents "no pain" and 10 represents "pain as bad as it could be". The patient will classify his pain during a complete isotonic unipodal squat on an inclined plane.
Pain intensity | Eigth weeks, before and after each intervention session
  This outcome will be evaluated by an 11-point scale ranging from 0 to 10, in which 0 represents "no pain" and 10 represents "pain as bad as it could be". The patient will rate the pain during rest before and after each intervention session.
Triple hop test | 8 weeks after randomization
  The patient will perform a test composed of three consecutive jumps, as far as possible, always landing on the same foot.
Pressure pain threshold | 8 weeks after randomization
  The patient will perform 10 repetitions of the complete unipodal squat on an inclined plane and sequentially will be placed on a stretcher lying comfortably with the knee flexed at 20 degrees. The patient should indicate the point of greatest pain in the tendon, which will be marked to be the location of the tip of the algometer, and the distance to the apex of the patella will be measured to use the same point in the assessment after treatment. If the patient does not present pain in the assessment after treatment, the point standardized in the initial evaluation will be used. If the patient still presents pain, the point of greatest pain will be evaluated. For measurement, pressure will be applied until the patient experiences a mild pain sensation (pain level 1), when he will be instructed to press the algometer button to stop the test.
Muscular strength | 8 weeks after randomization
  The hand dynamometer will be used to measure the strength of the quadriceps femoris, hamstring, gluteus maximus, gluteus medius and lateral hip rotators.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina MN Cabral, PhD, Principal Investigator — Universidade Cidade de São Paulo
Locations (1):
- Physical Therapy Outpatient Department, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No